CLINICAL TRIAL: NCT07286682
Title: A Phase 1, Randomized, Placebo-Controlled Single Ascending Dose Participant- and Investigator-Blind Study to Investigate the Safety, Tolerability, and Pharmacokinetics of UCB5285 in Healthy Study Participants
Brief Title: A Study to Investigate the Safety, Tolerability, and Pharmacokinetics of UCB5285 in Healthy Study Participants
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: UCB Biopharma SRL (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Basic Science
Other Study IDs: UP0161
Record Dates: First submitted 2025-12-03; First posted 2025-12-16 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Healthy Participants
Keywords: UCB5285

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Cohort 1 (Experimental): Participants randomized to this arm will receive a single dose of UCB5285 (Dose 1) or placebo via Route of Administration 1.
  Interventions: Drug: UCB5285; Other: Placebo
- Cohort 2 (Experimental): Participants randomized to this arm will receive a single dose of UCB5285 (Dose 2) or placebo via Route of Administration 1.
  Interventions: Drug: UCB5285; Other: Placebo
- Cohort 3 (Experimental): Participants randomized to this arm will receive a single dose of UCB5285 (Dose 3) or placebo via Route of Administration 1.
  Interventions: Drug: UCB5285; Other: Placebo
- Cohort 4 (Experimental): Participants randomized to this arm will receive a single dose of UCB5285 (Dose 4) or placebo via Route of Administration 1.
  Interventions: Drug: UCB5285; Other: Placebo
- Cohort 5 (Experimental): Participants randomized to this arm will receive a single dose of UCB5285 (Dose 4) or placebo Route of Administration 2.
  Interventions: Drug: UCB5285; Other: Placebo
- Cohort 6 (Experimental): Participants randomized to this arm will receive a single dose of UCB5285 (Dose 5) or placebo via Route of Administration 1.
  Interventions: Drug: UCB5285; Other: Placebo
- Cohort 7 (Experimental): Participants randomized to this arm will receive a single dose of UCB5285 (Dose 5) or placebo via Route of Administration 2.
  Interventions: Drug: UCB5285; Other: Placebo
- Cohort 8 (Experimental): Participants randomized to this arm will receive a single dose of UCB5285 (Dose 6) or placebo via Route of Administration 1.
  Interventions: Drug: UCB5285; Other: Placebo

INTERVENTIONS:
Drug: UCB5285 — Participants will receive UCB5285 as prespecified in each cohort.
Other: Placebo — Participants will receive matching placebo as prespecified in each cohort.

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of single ascending doses of UCB5285 in healthy study participants, including healthy Japanese study participants

ELIGIBILITY:
Inclusion Criteria:

* For study participants of Japanese origin: study participant who is born in Japan and of Japanese descent as evidenced in appearance and verbal confirmation of familial heritage with all 4 grandparents and both parents born in Japan and has not had a significant change in lifestyle or diet since leaving Japan
* For all study participants:
* Study participant must be 18 to 55 years of age, inclusive, at the time of signing the informed consent
* Study participants who are overtly healthy as determined by medical evaluation including medical history, physical examination, laboratory tests, and cardiac monitoring.
* Body weight within 40 kilograms (kg) to 110 kg and body mass index (BMI) within the range of 18 kilograms per meter square (kg/m2) to 30 kg/m2 (inclusive)

Exclusion Criteria:

* Study participant has a history or presence of any medical or psychiatric condition, physical examination finding, laboratory test result, electrocardiogram (ECG), or vital sign that, in the opinion of the investigator, could significantly alter the absorption, or elimination of drugs; constitute a risk when taking the study intervention; or interfere with the interpretation of data
* Study participant has a recent history (within 6 months of Screening) or currently active clinically significant bacterial, fungal, endoparasite, or viral infection.
* Study participant has a significant allergy to humanized monoclonal antibody (mAbs)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 96 (Estimated)
Dates: Start 2025-12-08 (Actual); Primary Completion 2026-12-13 (Estimated); Study Completion 2026-12-13 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events (TEAEs) | From Day 1 to the End Of Study (up to Day 161)
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. Treatment emergent adverse events (TEAEs) are adverse events that are not present prior to the pharmaceutical product administration or an already present event that worsens either in intensity or frequency.
Incidence of Treatment-Emergent Serious Adverse Events (SAEs) | From Day 1 to the End Of Study (up to Day 161)
  An SAE is defined as any untoward medical occurrence that, at any dose, meets 1 or more of the criteria listed:
  * Results in death
  * Is life-threatening
  * Requires inpatient hospitalization or prolongation of existing hospitalization
  * Results in persistent or significant disability/incapacity
  * Is a congenital anomaly/birth defect
  * Other important medical events which based on medical or scientific judgement may jeopardize the patients or may require medical or surgical intervention to prevent any of the above.

SECONDARY OUTCOMES:
Maximum Observed Serum Concentration (Cmax) of UCB5285 | From Day 1 (Predose) at predefined time points up to Day 161
  Maximum observed serum concentration (Cmax) of UCB5285
Area Under the Serum Concentration-Time Curve From Time Zero to Infinity (AUC) of UCB5285 | From Day 1 (Predose) at predefined time points up to Day 161
  Area under the serum concentration-time curve from time zero to infinity (AUC) of UCB5285
Area Under the Serum Concentration-Time Curve from Time Zero to the Time of Last Detectable Concentration (AUC0-t) of UCB5285 | From Day 1 (Predose) at predefined time points up to Day 161
  Area under the serum concentration-time curve from time zero to the time of last detectable concentration (AUC0-t) of UCB5285

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — 001 844 599 2273 (UCB)
Locations (1):
- Up0161 1001, Harrow, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Due to the small sample size in this trial, individual participant-level data cannot be adequately anonymized as there is a reasonable likelihood that individual participants could be re-identified. For this reason, data from this trial cannot be shared.